CLINICAL TRIAL: NCT07233057
Title: The Effect of Ice-Cold Mentholated Water Spray on Thirst Perception, Dry Mouth, Nausea, and Physiological Parameters in the Post-Rhinoplasty Period
Brief Title: The Effect of Ice Cold Mentholated Water Spray After Rhinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/11/01/4
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Rhinoplasty
Keywords: Ice water spray; Mentholated cold water spray

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ice water spray (Experimental)
  Interventions: Other: Ice water spray
- Menthol Cool Water Spray (Experimental)
  Interventions: Other: Menthol Cool Water Spray
- Control (No Intervention)

INTERVENTIONS:
Other: Menthol Cool Water Spray — Sterile ice water with menthol, cooled between 0-6°C in the refrigerator, will be stored in glass bottles with oral spray heads. The first application will be made half an hour after extubation, and then every hour for the next three hours. The spray will be applied to different areas of the patient's mouth (upper jaw, lower jaw, left cheek, right cheek, and tongue).
  Arms: Menthol Cool Water Spray
Other: Ice water spray — Sterile ice water, cooled to 0-6°C in the refrigerator, will be stored in glass bottles with oral spray heads. The first application will be made half an hour after extubation, and then every hour for the next three hours. The spray will be applied to different areas of the patient's mouth (upper jaw, lower jaw, left cheek, right cheek, and tongue).
  Arms: Ice water spray

SUMMARY:
This clinical trial aims to evaluate the effects of a menthol-infused cold water spray on thirst perception, dry mouth, nausea, and physiological parameters in patients after rhinoplasty. The intervention is expected to provide a refreshing sensation, alleviate discomfort associated with postoperative thirst and dryness, and contribute to improved patient comfort and recovery. Physiological parameters such as heart rate, blood pressure, and oxygen saturation will also be monitored to assess systemic effects.

ELIGIBILITY:
Inclusion Criteria:

* Must be extubated in the surgical intensive care unit after surgery for at least 3 hours or more
* Must be 18 years of age or older
* Must be conscious and oriented to time and place
* Must be ASA class I-III and Mallampati class I-II, must have a Mann assessment of swallowing ability score of ≥95, and must have a Glasgow Coma Scale (GCS) score of 15
* Must have given informed consent to participate in the study

Exclusion Criteria Patients were excluded from the study if they had: • Ingestion or absolute contraindications to swallowing any substance,

* Mandibular trauma,
* Patients undergoing ear, nose, and throat, intracranial, or oral surgery,
* Patients allergic to menthol or those who do not prefer menthol water,
* Patients with compromised oral and lingual mucosal integrity before surgery,
* Patients with any neurological, renal, cardiac, or pulmonary disease,
* Patients taking psychoactive medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Severity of dry mouth | The samples were evaluated at 4 time points: immediately before the first application (To) and 30 minutes after each of the three applications (T1, T2, T3).
  Severity of dry mouth The severity of dry mouth was assessed using a VAS with a score between 0 and 10 (0 = I do not experience dry mouth at all, 10 = I experience very severe dry mouth).
Nausea Severity | The samples were evaluated at 4 time points: immediately before the first application (To) and 30 minutes after each of the three applications (T1, T2, T3).
  Nausea is assessed in the same way using the Vas. Nausea is assessed by labeling one end of the scale as "no nausea" and the other as "very severe nausea" and asking the patient to place a mark on the scale indicating the severity of nausea. The distance (in cm) from the "no nausea" end of the scale to the mark made by the patient is used to measure the patient's nausea.
372 / 5.000 Thirst Severity | The samples were evaluated at 4 time points: immediately before the first application (To) and 30 minutes after each of the three applications (T1, T2, T3).
  A Visual Analog Scale (VAS) was used to assess the subjects' thirst severity, with a score ranging from 0 to 10 (0 = not at all, 10 = very severe).
Physiological Parameters Tracking Form | The samples were evaluated at 4 time points: immediately before the first application (To) and 30 minutes after each of the three applications (T1, T2, T3).
  This form was also developed by the researchers and included heart rate, systolic and diastolic blood pressures, and oxygen saturation levels. Participants' physiological parameters were recorded a total of four times in both groups: once at baseline and then 30 minutes after each exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)